CLINICAL TRIAL: NCT01208883
Title: A FEASIBILITY STUDY ON CONTINUOUS ADAPTIVE [18F]FDG-PET-GUIDED RADIOTHERAPY FOR HEAD AND NECK CANCER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010/510
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Squamous Cell Carcinoma
Keywords: Primary non-operated squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx and larynx.
MeSH Terms: conditions — Carcinoma, Squamous Cell; Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- repetitive per-treatment [18F]FDG-PET for treatment adaptation (Experimental)
  Interventions: Other: repetitive per-treatment [18F]FDG-PET for treatment adaptation

INTERVENTIONS:
Other: repetitive per-treatment [18F]FDG-PET for treatment adaptation — repetitive per-treatment [18F]FDG-PET for treatment adaptation

SUMMARY:
Treatment adaptation to biological and anatomical changes occurring during treatment can increase the chance of cure at minimized radiation-induced toxicity in head and neck cancer patients. This trial investigates the feasibility of using repetitive per-treatment [18F]FDG-PET acquired during treatment in adaptive [18F]FDG-PET-voxel intensity-based intensity-modulated radiotherapy (IMRT) or volumetric-modulated arc therapy (VMAT) for head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx.
* Primary unresectable tumor and/or patients refused surgery.
* Stage T1-4; T3-4 N0 or Tany N1-3 for cancer of the glottis.
* Multidisciplinary decision of curative radiotherapy or radiochemotherapy.
* Karnofsky performance status ≥70%.
* Age ≥ 18 years old.
* Informed consent obtained, signed and dated before specific protocol procedures.

Exclusion Criteria:

* Treatment combined with brachytherapy.
* Prior irradiation to the head and neck region.
* Distant metastases.
* Second primary tumors that are not under control
* Pregnant or lactating women.
* Creatinine clearance (Cockcroft-Gault) ≤ 60 mL/min before treatment.
* Allergy to the CT-contrast agents.
* Mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study.
* Patient unlikely to comply with protocol, i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To assess volume changes of the targets and organs at risk as detected by repetitive per-treatment [18F]FDG-PET/CT. | at time of per-treatment [18F]FDG-PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Neve, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website University Hospital Ghent, Belgium — http://www.uzgent.be